CLINICAL TRIAL: NCT06766617
Title: Assessment of Insulin Sensitivity in Healthy Adults by a 13C-glucose Breath Test : Method Development and Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 16.02.BIO
Record Dates: First submitted 2024-07-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Insulin Sensitivity/Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Monocentric, sequential open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucose 75 Gr (Experimental): 75g of anhydrous glucose dissolved in 375 ml of water (Vittel) mixed with 150mg of U-13C]-glucose (stable isotope from Eurisotope, France).
  Interventions: Other: 75 gr Glucose

INTERVENTIONS:
Other: 75 gr Glucose — 75g of anhydrous glucose dissolved in 375 ml of water (Vittel) mixed with 150mg of U-13C]-glucose (stable isotope from Eurisotope, France). will be orally taken
  Other Names: oral glucose intake

SUMMARY:
The current research project aims to assess the insulin resistance (less sensitivity), from measures of insulin and glucose in response to a standard oral intake of glucose (standardized oral glucose tolerance test). For this, we wish to test and validate the method of glucose labelled 13-C (stable isotope) breath test in comparison with standardized methods to measure glucose and insulin. Comparative methods that will be used are measures of glycemia from venous blood withdrawal and continuous glucose measurement in the skin tissue (external face of the arm) using the Abbott's freestyle libre system.

Repeatability and reliability of the 13-C glucose breath test will be checked from repeated measures over time.

DETAILED DESCRIPTION:
The current research project aims to assess the insulin resistance (less sensitivity), from measures of insulin and glucose in response to a standard oral intake of glucose (standardized oral glucose tolerance test). For this, we wish to test and validate the method of glucose labelled 13-C (stable isotope) breath test in comparison with standardized methods to measure glucose and insulin. Comparative methods that will be used are measures of glycemia from venous blood withdrawal and continuous glucose measurement in the skin tissue (external face of the arm) using the Abbott's freestyle libre system.

Repeatability and reliability of the 13-C glucose breath test will be checked from repeated measures over time.

ELIGIBILITY:
Inclusion Criteria:

Healthy male adults aged 18-40 Able to understand and to sign a written informed consent

Exclusion Criteria:

* EXCLUSION CRITERIA
* Known type 1 or type 2 diabetes, by anamnesis
* Family history of type 2 diabetes (parents)
* History of gestational diabetes
* Any other metabolic disease possibly impacting the postprandial glucose and insulin response (anamnesis)
* Any medication impacting the energetic metabolism, to the opinion of the investigator
* Pregnant or lactating women (anamnesis)
* Smoking
* Allergy or intolerance to any food or compound used in this study
* Currently following a strict exercise program (more than three times per week) in order to either lose weight, gain muscle or reach competition standards for a chosen sport
* Having given blood in the past three months or willing to give blood in the 3 months following the completion of the study
* Currently participating or having participated in another clinical trial during the past month.
* Volunteer who cannot be expected to comply with the protocol

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — excluded hormonal variability of young female participants
Enrollment: 7 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
1) To assess the within-subjects variability and overall repeatability of the 13C-glucose breath test | 0 to 300 minutes, after oral administration
  repeated measure of breath over the 3 visits.

SECONDARY OUTCOMES:
Compare the results of breath test and CGM with the classical indexes of insulin resistance after an oral glucose challenge (OGTT) containing a small amount of [U13C]-glucose. | 0 to 300 minutes, after oral adminstration
  repeated measure over the 3 visits of breath, plasma and CGM values
Repeatability of the continuous glucose monitoring system (CGM) | 0 to 300 minutes, after oral adminstration
  repeated measure over the 3 visits of breath, plasma and CGM values

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical innovation lab, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No
No sharing planned